CLINICAL TRIAL: NCT06574035
Title: Michigan Men's Diabetes Project 3 (MenD 3): Mind and Motion
Brief Title: Michigan Men's Diabetes Project III(MenDIII): Mind and Motion
Acronym: MenDIII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jaclynn Hawkins, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00256519
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2; Depressive Symptoms; Depression
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression | interventions — Cognitive Behavioral Therapy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants randomized to the intervention group will receive 8 one hour virtual sessions of individual cognitive behavioral therapy (CBT) that will take place via U-M Zoom, which is a HIPAA compliant virtual conferencing platform.
  Participants in this group will also receive 8 one hour virtual sessions of individual exercise.
  Participants in this group will also receive 8 one hour virtual group discussion sessions that will serve as on-going support. This group (4-8 participants) discussion will be facilitated by one CBT Interventionist and one Exercise Interventionist. These sessions will take place following the individual sessions of CBT and Exercise.
  Interventions: Behavioral: Cognitive Behavioral Therapy; Behavioral: Exercise; Behavioral: Group Discussions - Ongoing Support
- Control Group (Active Comparator): Participants randomized to the control group will receive enhanced usual care (EUC). The EUC group will receive 8 sessions of standard Cognitive Behavioral Therapy.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive behavioral therapy focuses on the unique needs of men. A culturally adapted CBT program will be administered to participants as it has demonstrated increased effectiveness for marginalized populations. Cognitive Behavioral Therapy (CBT) aligns well with these cultural needs due to its individualized approach, non-judgmental stance, collaborative nature, and emphasis on empowerment through skills building.
Behavioral: Exercise — Research demonstrates a preference for physical activity interventions among men with chronic illnesses, while highlighting limited access to fitness facilities in low-income urban areas as a barrier to participation. Online physical activity interventions have shown efficacy and cost-effectiveness in improving health behaviors, with virtual exercise programs for low-income African American populations demonstrating significant reductions in depressive symptoms. Therefore participants will receive exercise to help improve their diabetes self-management behaviors and depressive symptoms.
  Arms: Intervention Group
Behavioral: Group Discussions - Ongoing Support — Participants will join group discussions that will serve as on-going support. The small group component is designed to foster self-efficacy, autonomous motivation, and enjoyment by integrating skills building, personal values, spirituality, and goal setting. This approach has shown positive outcomes in previous pilot studies with African American men, serving as a source of vicarious learning and social support.
  Arms: Intervention Group

SUMMARY:
The Michigan Men's Diabetes Project III: Mind & Motion is an 7-month pilot randomized clinical trial. The investigators are looking to recruit 80 Black men with type 2 diabetes (T2D) (need to have diagnosis for at least one year) that are over the age of 18. Participants also must be under the care of a physician for their diabetes, self report an Hemoglobin A1c (A1C) of 7.0% or more in the last year, be willing to participate in study events (weekly physical activity, exercise and Cognitive Behavioral Therapy (CBT) sessions, group discussion sessions, and in-person health assessments), have reliable internet access (steady internet connection or unlimited data) that will allow them to use a tablet/phone/computer to complete study related tasks, live in the Wayne or Washtenaw County, and have reliable transportation to in-person events. All participants will receive 8 hours/sessions of cognitive behavioral therapy. Participants randomized to the intervention arm will also receive 8 sessions of guided exercise at the same time. Following that they will also receive 8 group discussion sessions that will serve as on-going support. All sessions will be help via Zoom. Additionally, all participants will participate in The 4 health assessments will take place at baseline, 10 weeks, 18 weeks, and 30 weeks.

ELIGIBILITY:
Inclusion Criteria:

* African American/Black males
* age 18 years or older
* ambulatory status
* diagnosis of Type 2 Diabetes (T2D) for one year duration or longer
* be under the care of a physician for their diabetes, self report an A1C of 7.0% or more in the last year
* be willing to participate in study events (weekly physical activity, exercise and CBT sessions, group discussion sessions, and in-person health assessments)
* have reliable internet access (steady internet connection or unlimited data) that will allow them to use a tablet/phone/computer to complete study related tasks
* live in the Wayne or Washtenaw County\
* have reliable transportation to in-person events

Exclusion Criteria:

* stage 2 hypertension as defined by Joint National Committee (JNC) VIII
* recent cardiac events
* recent laser surgery for proliferative retinopathy
* history of stroke
* lower limb amputation
* peripheral neuropathy
* severe Chronic Obstructive Pulmonary Disease (COPD) (e.g., basal oxygen)
* class III or IV heart failure
* medical instability.

Per American College of Sports Medicine (ACSM) guidelines, medical exclusion criteria will also include currently experiencing:

* ongoing unstable angina
* uncontrolled cardiac arrhythmia with hemodynamic compromise
* active endocarditis
* symptomatic severe aortic stenosis
* acute myocarditis or pericarditis
* acute aortic dissection
* acute pulmonary embolism
* pulmonary infarction
* deep venous thrombosis
* physical disability that precludes safe and adequate testing
* chest discomfort with exertion
* unreasonable breathlessness, or dizziness, fainting, or blackouts.

As part of the screening process, the investigators will ask the participant to self-report on these conditions. Participants who are currently receiving psychotherapy services for the treatment of depression from a mental health provider will be excluded. Participants who are currently receiving only medication management from a psychiatrist will be included.

If you are interested in the study, please complete our screening survey: https://redcapproduction.umms.med.umich.edu/surveys/?s=JNPPEDANX7KLPPF9. Thank you so much!

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation of gender identity
Enrollment: 80 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in A1C | Screening, Baseline, 10 weeks, 18 weeks, 30 weeks
  Anthropometric/clinical data
Change in General Quality of Life (12-Item Short Form Survey (SF-12)) | Baseline, 10 weeks, 18 weeks, 30 weeks
  Survey Data - 12 questions covering physical and mental health domains - Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.
Change in Diabetes-Related Distress (The Type 2 Diabetes Distress Assessment System) | Baseline, 10 weeks, 18 weeks, 30 weeks
  Survey Data - The assessment system has two components: The Core Distress Scale and The Sources Scale. The CORE DISTRESS SCORE is simply the average of the 8 items of the CORE SCALE, with each item rated on a 1 to 5 scale: Mean score < 2.0 indicate little or no distress, Mean score between 2.0 and 2.9 indicate moderate distress, Mean score > 3.0 indicate high distress. The Sources scale aims to find the sources of the distress, whether CORE DISTRESS is high or low, it is helpful to identify those aspects of living with diabetes that are contributing to the individual's diabetes distress.
Change in Diabetes Quality of Life (Diabetes Quality of Life Instrument) | Baseline, 10 weeks, 18 weeks, 30 weeks
  Survey Data - Survey answers range for each section of the survey asking about satisfaction, worry, and impact of diabetes. The DQoL measure consists of 46 items ranked on a 5-point Likert scale. Individual domain and DQoL total scores range from 0 (lowest possible QoL) to 100 (highest possible QoL).

SECONDARY OUTCOMES:
Change in Diabetes Self-Efficacy (Perceived Diabetes Self-Management Scale) | Baseline, 10 weeks, 18 weeks, 30 weeks
  Survey Data - The scale is an 8-item scale that uses a 5-point Likert scale to measure self-efficacy in diabetes management. The scale ranges from 8 to 40 points, with higher scores indicating greater self-efficacy.

OTHER OUTCOMES:
Change in Masculinity Ideology (The Conformity to Masculine Norms Inventory-30) | Baseline, 10 weeks, 18 weeks, 30 weeks
  Survey Data - The CMNI-30's subscales are scored by adding up the scores of each item. It is a 30-item scale that measures how much a person conforms to masculine norms in US society. The items are rated on a six-point Likert scale, ranging from 0 (strongly disagree) to 5 (strongly agree), with nine items reverse-coded.
Change in BMI | Baseline, 10 weeks, 18 weeks, 30 weeks
  Anthropometric/clinical data
Chance in Estimated Abdominal Subcutaneous and Visceral Fat Stores | Baseline, 10 weeks, 18 weeks, 30 weeks
  Anthropometric/clinical data
Change in Diabetes Social Support (Duke/UNC Functional Social Support) | Baseline, 10 weeks, 18 weeks, 30 weeks
  Survey Data - Responses are scaled on a 1-5 scale and tallied to create a total score with higher values indicating greater social support.
Sociodemographic characteristics | Baseline
  Survey Data
Healthcare utilization | Baseline
  Survey Data
Comorbidities | Baseline
  Survey Data
Change in Medication Adherence (Adherence to Refills and Medicines Scale for Diabetes) | Baseline, 10 weeks, 18 weeks, 30 weeks
  Survey Data - The scale a 14-question survey that measures self-reported medication adherence. The ARMS-D is designed to be brief and easy to use, and can help identify reasons for non-adherence. Each item on the scale is rated on a four-point Likert scale, with 1 being "none of the time" and 4 being "all of the time". The items are then summed to create a score that ranges from 11 to 44, with higher scores indicating better adherence.
Change in Aerobic Capacity (6 minute walk test) | Baseline, 10 weeks, 30 weeks
  Anthropometric/clinical data
Change in Working Alliance between Counselor & Participant (Working Alliance Inventory - Short Revised) | Up to 8 weeks
  Survey Data - The Scale is 12 questions, Each item is scored from 1-7, minimum=1 to maximum=7, ranging from Never to Always. Higher scores reflect a more positive rating of working alliance.
Change in Metabolic Control (continuous blood glucose levels) | Up to 18 weeks
  Anthropometric/clinical data
Change in Depression Symptoms (Patient Health Questionnaire 9) | Screening and throughout study completion, up to 30 weeks.
  Survey Data - Answer Options rang from Not at all = 0, Several days = 1, More than half the days = 2, Nearly every day = 3. Scores can range from 1 - 27, the higher the score, the more severe the depression.
Change in Blood Pressure (systolic and diastolic) | Baseline, 10 weeks, 18 weeks, 30 weeks
  Anthropometric/clinical data
Change in Physical Activity Regimen | Up to 18 weeks
  Exercise Log Data
Change in Heart Rate | Baseline, 10 weeks, 18 weeks, 30 weeks
  Anthropometric/clinical data

CONTACTS AND LOCATIONS:
Overall Officials: Jaclynn Hawkins, PhD, Principal Investigator — University of Michigan, School of Social Work
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States